CLINICAL TRIAL: NCT05688462
Title: Studying Trends of Auto-Regulation in Severe Head Injury in Paediatrics
Acronym: STARSHIP
Status: Completed | Type: Observational
Sponsor: Shruti Agrawal (Other)
Collaborators: Action Medical Research (Other)
Responsible Party: Sponsor-Investigator, Shruti Agrawal, Consultant PIC, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Other Study IDs: ADDENBROOKESHPTBI
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: TBI (Traumatic Brain Injury)
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data Collection — This is an observational prospective cohort study. Children admitted to ten identified PICUs in the UK with severe TBI with a clinical need for ICP and ABP monitoring will be included for data collection. The database will contain routinely monitored physiological parameters during management of PTBI in PICU. Without disturbing the routine care and management of these patients, investigators aim to collect this data continuously in a bedside laptop equipped with the study software (ICM+, Cambridge Enterprise Ltd, Cambridge, UK). Alongside these physiological parameters, investigators will also collect relevant clinical and demographic data (details below) and follow these patients for up to 12 months post ictus to assess neuro-psychological outcome.

SUMMARY:
Children are known to have devastating impact from traumatic brain injury (TBI). The focus of treatment of severe TBI is to limit secondary insult which can aggravate brain injury and worsen outcome and is supported by monitoring brain pressure (ICP) and arterial pressure (ABP). These pressures, if incorporated in Multi-modality monitoring can be used to interpret state of mechanisms used by brain to maintain normal blood flow. This has been advised to guide management of severe TBI in adults, however, there is limited experience with advanced brain monitoring in children. The investigators propose to study the use of this in children with severe TBI. Children (up to 16 years of age) with a severe TBI are referred to a neurosurgical unit (NSU) and admitted to a paediatric intensive care unit (PICU) as part of usual NHS clinical practice. All patients with a severe TBI require a monitoring wire to be inserted into the brain to read the pressure inside the skull and a similar device in an artery to monitor the blood pressure. These recordings are documented by a PICU nurse at a prescribed frequency. Without interrupting this clinical practice investigators propose to record these values using computer software called ICM+. These recordings will provide real time analysis and a continual recording of important parameters which will provide the study with much needed information on the patterns of pressures in the brain after this injury in children. All patients will be followed up for 12 months to see how well they recover, neuropsychology assessment will be performed by a Neuropsychologist at the recruiting centre using a standardised form.

DETAILED DESCRIPTION:
This is an observational prospective cohort study. Children admitted to ten identified PICUs in the UK with severe TBI with a clinical need for ICP and ABP monitoring are being included for data collection. The database will contain routinely monitored physiological parameters during management of PTBI in PICU. Without disturbing the routine care and management of these patients, investigators are collecting this data continuously in a bedside laptop equipped with the study software (ICM+, Cambridge Enterprise Ltd, Cambridge, UK). Alongside these physiological parameters, investigators are also collecting relevant clinical and demographic data (details below) and follow these patients for up to 12 months post ictus to assess neuro-psychological outcome. The created database will be used to analyze the state of cerebral autoregulation. Investigators will also analyze the data to see if investigators can derive optimal cerebral perfusion pressures based on the state of autoregulation and compare it with the patient outcome at 6 and 12 months. The database can also be subsequently used in the future projects testing hypotheses inspired by the experience gained in the adult TBI population research & to answer important questions about severe PTBI.

Inclusion Criteria:

* Patients 16 years old or younger at the time of injury
* Admitted to PICU for management of TBI
* TBI-related pathology confirmed on CT or MRI
* Clinical requirement for invasive monitoring of ICP and ABP

Exclusion Criteria:

- None

Study Aim: The investigators aim to create a research database of high-resolution monitoring data from PTBI patients along with the clinical and demographic details and neuro-psychological outcome up to 12 months post-ictus, from 10 UK PICUs to be used for research purposes. As the first step, investigators analyze the data to determine retrospective optimal clinical parameters when managing these patients. The investigator's hypothesis is that investigators can define the optimal parameters for CPP based on indices of autoregulation (PRx) and that the optimal parameters of CPP and PRx in PTBI will differ to adults, both qualitatively and quantitatively.

Study Objectives:

Primary Objective: To detect thresholds of PRx associated with favourable outcome in PTBI.

Secondary objectives:

1. Characterise patterns of optimal CPP in PTBI as a function of age, severity and character of injury, intracranial pressure, etc.
2. Compare the fluctuations in these measured parameters with the outcome.
3. Establish a comprehensive paediatric database of a basic set of high resolution (pulse waveforms resolution) neuro-monitoring data including ICP, ABP and ECG.

Patient Recruitment and Consent: Each PTBI patient admitted to the recruiting PICU with invasive monitoring of ICP and ABP is considered for recruitment. The research team at each recruiting PICU identifies the patients and sets up high-resolution data collection to the project laptop under an anonymised ID as soon as possible after the patient has been commenced on invasive monitoring and stabilized on PICU. Physiological and clinical data is recorded under this unique study ID. As the acute phase of the project is purely observational and does not involve any therapeutic intervention or change in regular standard care, investigators take a deferred consent for acute data collection and sharing. This is important to obtain a bias-free sample and ensure capture of early changes in intracranial physiology after head injury. When appropriate, the identified guardian/parent is informed and consented for data sharing and follow-up before the patient is discharged from the hospital. For patients who die before the consent can be obtained, the clinician in charge of patient's clinical care only (not study team) will access and anonymise data of the deceased patient under his/her clinical care; this anonymised data will then be provided to the study team.

Data Collection: ICP is monitored with an intraparenchymal microsensor inserted into the right (predominately but can be left) frontal cortex and ABP is monitored in the radial or femoral artery with a zero calibration at the level of the right atrium. The head end elevation is part of the standard international protocol for management for PTBI, and any deviations from this policy in individual cases will be recorded. Full resolution data of routinely monitored physiological parameters in managing PTBI [ICP, ABP, ETCO2, SpO2 and ECG] is collected from bed-side monitors. Pulsatile signals [ICP, ABP and ECG] are recorded with the maximum sampling frequency offered by the bed-side monitors, at least 100 Hz for invasive pressures, and at least 200Hz for ECG. This is done using relevant, monitor type specific, data export protocols implemented in the study (ICM+) software running on a bed-side laptop. The same software will be later used for the retrospective analysis of all stored signals. The continuous data collection is stopped when the patient either starts to wake up or dies and the invasive monitoring is stopped. Apart from general demographics and clinical data, the other data being collected are mechanism and details of injury, relevant past history, post resuscitation Glasgow coma scale, initial pupillary size and reactivity, pre-hospital hypoxia/ hypotension/ hyperthermia/ cardiopulmonary resuscitation, injury & disease severity scores (Pediatric Index of Mortality- PIM II score, Injury Severity Score- ISS), CT scan findings. The investigators are also collecting: daily laboratory values (hemoglobin, glucose, sodium, lactate), PaO2, PaCO2 and FiO2, PEEP, medical interventions for TBI (positioning, collar, temperature, CO2, glucose, hypertonic saline or mannitol, sedation/paralysis, barbiturate coma, anti-seizure medication, use of vasoactive drugs to maintain blood pressure & surgical interventions (haematoma evacuation, elevation of depressed fracture, CSF diversion-external ventricular drainage, new brain imaging, any other relevant event.

ELIGIBILITY:
Inclusion Criteria:

* Patients 16 years old or younger at the time of injury
* Admitted to PICU for management of TBI
* TBI-related pathology confirmed on CT or MRI
* Clinical requirement for invasive monitoring of ICP and ABP

Exclusion Criteria:

- None

Ages: 3 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children upto the age of 16 years with TBI identified on CT/MRI with a clinical need for invasive blood pressure and intracranial pressure monitoring
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
To detect thresholds of PRx associated with favourable outcome in PTBI | 12 months

SECONDARY OUTCOMES:
Characterise patterns of optimal CPP in PTBI as a function of age, severity and character of injury, intracranial pressure | 12 months
Compare the fluctuations in these measured parameters with the outcome. | 12 months
Establish a comprehensive paediatric database of a basic set of high resolution (pulse waveforms resolution) neuro-monitoring data including ICP, ABP and ECG | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Shruti Agrawal, MD, Principal Investigator — Cambridge University Hospitals Nhs Foundation Trust - Cambridge, Cambridgeshire
Locations (1):
- Shruti Agrawal, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
On request. Data to be stored in a non-public secure reporsitory

REFERENCES:
- [Background] Agrawal S, Smith C, Bogli SY, Placek MM, Cabeleira M, White D, Daubney E, Young A, Beqiri E, Kayani R, O'Donnell D, Pathan N, Watson S, Maw A, Ganrett M, Kanthimathinathan HK, Bangalore H, Sundararajan S, Subramanian G, Raffaj D, Sarfatti A, Lampareillo S, Mayer A, Ross O, Czosnyka M, Hutchinson PJ, Smielewski P; STARSHIP study team. Status of cerebrovascular autoregulation relates to outcome in severe paediatric head injury: STARSHIP, a prospective multicentre validation study. EClinicalMedicine. 2025 Feb 5;81:103077. doi: 10.1016/j.eclinm.2025.103077. eCollection 2025 Mar. PMID 39996125
- [Derived] Agrawal S, Placek MM, White D, Daubney E, Cabeleira M, Smielewski P, Czosnyka M, Young A, Watson S, Maw A, Hutchinson PJ. Studying Trends of Auto-Regulation in Severe Head Injury in Paediatrics (STARSHIP): protocol to study cerebral autoregulation in a prospective multicentre observational research database study. BMJ Open. 2023 Mar 10;13(3):e071800. doi: 10.1136/bmjopen-2023-071800. PMID 36898758